CLINICAL TRIAL: NCT03834480
Title: Ultra Sound Guided Injection of Platelet Rich Plasma Versus Steroid for Sacroiliac Joint Pain
Brief Title: Intraartecular Platelet Rich Plasma for Sacroiliitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS17.10.03
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Sacroiliitis
Keywords: Platelet reach plasma; sacroiliac; Ultrasound; Steroid; Chronic low back Pain
MeSH Terms: conditions — Sacroiliitis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • Steroid Group (S) (Experimental)
  Interventions: Other: Ultrasound guided Sacroiliac intra-articular injection
- • Platelet rich plasma Group (PRP) (Experimental)
  Interventions: Other: Ultrasound guided Sacroiliac intra-articular injection

INTERVENTIONS:
Other: Ultrasound guided Sacroiliac intra-articular injection — At the level of the sacral hiatus, the sacral cornuae were identified. posterior aspect of the sacroiliac joint, at 4.5 cm depth the SIJ was found. localal anesthetic was injected at the medial edge of the transducer, the spinal needle was advanced in a medial to lateral direction, under direct vision, until the needle was positioned in the SIJ. Local steroid solution or PRP 4ml volume was injected according to the study group and patient enrollment. If the injection is extra-articular, injectate (hyperechoic solution as it contains particulate steroid) can be seen spreading medially over the sacrum. The visual analog score, Oswestry Disability Index (ODI) score and the overall success rate basal, after one week,after one month,after three and six month's follow-up period after the initial block.

SUMMARY:
Comparison between the effect of steroids and platelet-rich plasma on low back pain after ultrasound-guided sacroiliac injection to determine any is more effective and of long duration

DETAILED DESCRIPTION:
A prospective randomized controlled study was conducted at the department of anesthesiology Mansoura University Hospital during the period from December 2017 to January 2019 on fifty ASA I-III adult patients, of both sex after approval of IRB (Institutional Review Board) ID number MS17.10.03 & IRB date 12-11-2017. The patients were randomly allocated into two groups each of 25 patients according to computer-generated random number codes that were placed in sealed envelopes, double blinded, with parallel-group comparison.

Steroid Group (S) (n. 25):- Patients were injected by 4 ml of sterile water containing the methylprednisolone Acetate (Depo-Medrol) per-kg calculated dose (0.5mg/kg up to a lean muscle body weight of 80kg in the painful sacroiliac joint).

Platelet rich plasma Group (P) (n. 25):-Patients received fixed volume of 4 ml platelet-rich plasma in the inflamed painful sacroiliac joint.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients of either sex. 2. ASA I&III. 3. Age between 18 - 70 years. 4. Chronic lower back pain of sacroiliac origin. 5. Anatomy of the joint can identified by the ultrasonography. Exclusion criteria

  1. Patients with contraindications to sacroiliac injection.
  2. Patients known to be allergic to platelet rich plasma or local anesthetics.
  3. History of immune suppression or immune compromised diseases
  4. Patient below age of 18 as the joint will undergo normal physiological changes.
  5. Patient over 70 years.
  6. Sacroiliac pain of multiple sources.
  7. Preoperative shivering or fever (>38oc).
  8. Hepatic, renal and heart failure patients.
  9. Patients on; anticoagulants, antiplatelet, and with INR≥1.5.
  10. Exclude corticosteroid injection in the sacroiliac joint at the last three months.
  11. Patient refusal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
visual analog score | Basal and after 6 months
  To evaluate the changes in visual analogue score over a 6-month follow-up period after intra-articular injection and compare these changes among the studied groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt